CLINICAL TRIAL: NCT04675099
Title: Promoting Caregiver-child Attachment and Recovery Through Early Intervention (pCARE): A Pilot Randomized Control Trial
Acronym: pCARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baystate Medical Center (Other)
Responsible Party: Principal Investigator, Elizabeth Peacock-Chambers, MD, Assistant Professor, Baystate Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: BH-20-132
Record Dates: First submitted 2020-11-18; First posted 2020-12-19 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Opioid-use Disorder; Substance Use Disorders; Parenting
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Standard Early Intervention services
  Interventions: Other: Standard Early Intervention services
- Intervention (Experimental): pCARE
  Interventions: Behavioral: pCARE; Other: Standard Early Intervention services

INTERVENTIONS:
Behavioral: pCARE — "Mothering from the Inside Out" is an evidence-based intervention delivered in substance use treatment settings that helps mothers with substance use disorders foster parent-child attachment, cope with stressful parenting situations, and promote their child's healthy development. This 3 month counseling intervention both improves parent-child attachment and decreases rates of drug relapse among mothers. The proposed mechanism of action targeted by the intervention is a change in parental reflective functioning, defined as the capacity to recognize and make sense of mental states (especially emotional states) and understand how they influence behavior and relationships.
  Other Names: Mothering from the Inside Out
  Arms: Intervention
Other: Standard Early Intervention services — The state of Massachusetts provides voluntary early childhood development services to substance-exposed infants through a system of Early Intervention programs. These programs offer coordinated services to all infants and toddlers with disabilities and those at risk for developmental delays in homes and child centers beginning at birth.

SUMMARY:
This purpose of this study is to use the existing infrastructure and therapeutic relationships developed by Early Intervention, a national system of child development programs, to make an evidence-based intervention for parents with substance use disorder, Mothering from the Inside Out, more readily accessible to postpartum women with substance use disorder. This study will assess the feasibility, acceptability, and preliminary outcomes of the intervention in a pilot randomized controlled trial. We will also identify key implementation domains that impact successful delivery. We hypothesize that the intervention will be feasible and acceptable to the study participants.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* 18 years of age or older
* Mother to an index child between birth and 2 years old at the time of estimated start of intervention delivery
* Engaged in formal recovery supports (including but not limited to: Recovery Coaches, support groups specific to people in recovery, medication assisted treatment) at time of enrollment for a minimum 3 months
* Willing to receive parenting supports for the index child through EI
* Geographically based within the catchment area of participating EI programs

Exclusion Criteria:

* Severe mental health problems (suicidal, homicidal, psychosis episodes within the past year)
* Significant cognitive impairment (unable to give informed consent)
* Has an index child that has complex medical problems that significantly impact the child's ability to interact with the parent (e.g. blindness, deafness, severe weakness, or paralysis)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-12-18 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Recruitment and enrollment | Through study completion up to 3 months
  The number of mothers referred, approached, and enrolled in the study
Number of Early Intervention services received | Through intervention period, an average of 6 months
  All Early Intervention services received by mothers and their child(ren)
The duration of intervention sessions | Through intervention period, an average of 6 months
  Session duration in minutes
The number of intervention sessions completed by mothers | Through intervention period, an average of 6 months
  The total number of sessions completed
Mothers' perceived barriers and facilitators to intervention delivery | Through intervention period, an average of 6 months
  Qualitative perceptions of intervention logistics
The number of supervision sessions completed by providers | Through intervention period for each mother participant, an average of 6 months
  The total number of sessions completed
Early Intervention and additional services received by mothers after intervention period | Post-intervention up to 3 months
  Services received qualitatively listed by mothers
Retention of study participants | Through study completion up to 3 months
  Time to loss of follow-up and perceived reason for discontinuation
Qualitative perceptions of intervention sessions from mothers | Through intervention period, an average of 6 months
  Open-ended feedback of intervention sessions
Qualitative perceptions of intervention sessions from Early Intervention providers | Through intervention period for each mother participant, an average of 6 months
  Open-ended feedback of intervention sessions
Qualitative perceptions of intervention sessions from Early Intervention providers after intervention period | Post-intervention for each mother participant up to 3 months
  Open-ended feedback via a 30-minute interview
Qualitative perceptions of intervention sessions from mothers after intervention period | 3 months after the completion of the intervention
  Open-ended feedback via a 30-minute interview
Adherence of providers to the intervention according to a revised 9-point "Mothering from the Inside Out" Adherence Rating Scale | Through intervention period for each mother participant, an average of 6 months
  The revised Mothering from the Inside Out (MIO) Adherence Rating Scale is a 9-item measure rated on a 3-point scale for frequency of occurrence (never or seldom, sporadically, or consistent) and competence (poorly executed, adequately executed, or well-executed) of intervention delivery. The measure uses intervention session audio- or video- recordings and includes MIO specific fidelity and a measure of therapeutic alliance.

SECONDARY OUTCOMES:
Changes in parental reflective functioning according to the Parent Development Interview (PDI) | 0, 3, and 6 months
  The Parent Development Interview (PDI) is a 14-item measure of parental reflective functioning in an interview format. Audio-recorded interviews are transcribed and coded on a 9-point Likert scale.
Changes in parent-child interactions according to the Coding Interactive Behavior (CIB) manual | 0, 3, 6 months
  Conducting a Free Play Session (a 10 minute video-recorded and coded interaction, face-to-face interaction (infants) or play session) and analyzing using 5-point Likert scale and the Coding Interactive Behavior (CIB) manual, a global coding system with 43 items (22 parent, 16 infant, and 5 dyadic codes). There are six composite scales for: maternal sensitivity, maternal intrusiveness, child involvement, child negative emotionality, dyadic reciprocity and dyadic negative states; and two additional constructs for 12-36 month olds: maternal limit setting and child compliance.

OTHER OUTCOMES:
Changes in psychiatric symptoms according to the Brief Symptom Index (BSI) | 0, 1, 2, 3, and 6 months
  The Brief Symptom Index (BSI) is a 53-item measure of psychiatric symptoms scored on a 5-point Likert scale (Cronbach's alpha = .97).
Changes in depressive symptoms according to the Patient Health Questionnaire-9 (PHQ-9) | 0, 1, 2, 3, and 6 months
  The Patient Health Questionnaire-9 (PHQ-9) is a widely used 9-item questionnaire rated on a 4-point scale with good psychometric properties including high internal consistency and construct validity.
Changes in substance use behavior according to the Addiction and Child Welfare Questionnaire (ACWQ) | 0, 1, 2, 3, and 6 months
  The Addiction and Child Welfare Questionnaire (ACWQ) assesses past substance use and involvement with child welfare systems with yes or no questions as well as frequency on a 4- or 5- point scale.
Changes in parenting stress according to the Parenting Stress Index (PSI) | 0, 1, 2, 3, and 6 months
  The Parenting Stress Index - Short Form (PSI) is a validated instrument assessing parenting stress (Cronbach's alpha = 0.93, test-retest coefficient = .96).
Child development using the Batelle Developmental Inventory | At baseline
  Batelle Developmental Inventory contains data collected as part of Early Intervention assessments per the Early Intervention evaluation schedule. All assessments collected during the enrollment period.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Peacock-Chambers, MD, MSc, Principal Investigator — Baystate Medical Center
Locations (1):
- Baystate Medical Center, Springfield, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No